CLINICAL TRIAL: NCT03984422
Title: Development of an Application for the Monitoring and Evaluation of Raynaud's Phenomenon
Brief Title: Application for Monitoring and Evaluation of Raynaud's Phenomenon
Acronym: RaynaudMoni
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.099; 2019-A00987-50 (Other: ID RCB)
Record Dates: First submitted 2019-05-24; First posted 2019-06-13 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Raynaud Phenomenon
Keywords: smartphone application; monitoring
MeSH Terms: conditions — Raynaud Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Raynaud phenomenon: Use of smartphone application
  Interventions: Other: Smartphone application

INTERVENTIONS:
Other: Smartphone application — use of smartphone application during 2 weeks to 3 months to collect frequency and duration of crises, RCS, photography of finger.

SUMMARY:
To evaluate the feasibility of using a smartphone application for monitoring and evaluation of Raynaud's Phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* primary or secondary Raynaud phenomenon clinically diagnosed by a physician
* Phone compatible with the application (most Android smartphones)
* Non-opposition of participation in the study
* Affiliation to the social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* Subject under administrative or judicial supervision
* Subject not speaking and not understanding French

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected in conjunction with a scheduled consultation in the Vascular Medicine Department or at the Clinical Research Center
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-03-31 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Satisfaction assessed by a 5-points Likert scales about using the application for the monitoring and evaluation of Raynaud's Phenomenon | 2 weeks
  The questionnaire assesses different items such as the ease of use of the application, the installation process on the smartphone, the use of reminders, etc. Overall satisfaction will be calculated as the non-weighted average of all items.

SECONDARY OUTCOMES:
Relationship between cutaneous digital temperature assessed by thermography and the severity of Raynaud's Phenomenon | 2 weeks
  Correlation between digital temperature and Raynaud's Condition Score (RCS)
Relationship between cutaneous digital temperature assessed by thermography and the frequency of RP attacks | 2 weeks
  Correlation between digital temperature and the daily frequency of attacks
Relationship between cutaneous digital temperature assessed by thermography and the duration of RP attacks | 2 weeks
  Correlation between digital temperature and the cumulative daily duration of attacks
Relationship between cutaneous digital temperature assessed by thermography and pain during RP attacks | 2 weeks
  Correlation between digital temperature and pain during attacks (assessed through a 10-point VAS)
Effect of Raynaud etiology on thermographic data | 2 weeks
  Comparison of cutaneous digital temperature between patients with primary and secondary Raynaud
Effect of Raynaud treatment on thermographic data | 2 weeks
  Comparison of cutaneous digital temperature between patients treated with calcium channel blockers and untreated patients

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Roustit, PharmD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Chu Grenoble Alpes, Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wigley FM, Flavahan NA. Raynaud's Phenomenon. N Engl J Med. 2016 Aug 11;375(6):556-65. doi: 10.1056/NEJMra1507638. No abstract available. PMID 27509103
- [Background] Herrick AL. The pathogenesis, diagnosis and treatment of Raynaud phenomenon. Nat Rev Rheumatol. 2012 Aug;8(8):469-79. doi: 10.1038/nrrheum.2012.96. Epub 2012 Jul 10. PMID 22782008
- [Background] Seibold JR, Wigley FM. Editorial: Clinical Trials in Raynaud's Phenomenon: A Spoonful of Sugar (Pill) Makes the Medicine Go Down (in Flames). Arthritis Rheumatol. 2017 Dec;69(12):2256-2258. doi: 10.1002/art.40307. Epub 2017 Nov 10. No abstract available. PMID 28859256
- [Background] Roustit M, Giai J, Gaget O, Khouri C, Mouhib M, Lotito A, Blaise S, Seinturier C, Subtil F, Paris A, Cracowski C, Imbert B, Carpentier P, Vohra S, Cracowski JL. On-Demand Sildenafil as a Treatment for Raynaud Phenomenon: A Series of n-of-1 Trials. Ann Intern Med. 2018 Nov 20;169(10):694-703. doi: 10.7326/M18-0517. Epub 2018 Oct 30. PMID 30383134
- [Background] Fava A, Wung PK, Wigley FM, Hummers LK, Daya NR, Ghazarian SR, Boin F. Efficacy of Rho kinase inhibitor fasudil in secondary Raynaud's phenomenon. Arthritis Care Res (Hoboken). 2012 Jun;64(6):925-9. doi: 10.1002/acr.21622. Epub 2012 Jan 24. PMID 22275160
- [Background] Denton CP, Hachulla E, Riemekasten G, Schwarting A, Frenoux JM, Frey A, Le Brun FO, Herrick AL; Raynaud Study Investigators. Efficacy and Safety of Selexipag in Adults With Raynaud's Phenomenon Secondary to Systemic Sclerosis: A Randomized, Placebo-Controlled, Phase II Study. Arthritis Rheumatol. 2017 Dec;69(12):2370-2379. doi: 10.1002/art.40242. PMID 29193819
- [Background] Maricq HR, Carpentier PH, Weinrich MC, Keil JE, Franco A, Drouet P, Poncot OC, Maines MV. Geographic variation in the prevalence of Raynaud's phenomenon: Charleston, SC, USA, vs Tarentaise, Savoie, France. J Rheumatol. 1993 Jan;20(1):70-6. PMID 8441170